CLINICAL TRIAL: NCT01867411
Title: Multimodal Neuroimaging Genetic Biomarkers of Nicotine Addiction Severity
Brief Title: Multimodal Neuroimaging Genetic Biomarkers of Nicotine AddictionSeverity
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913485; 13-DA-N485
Record Dates: First submitted 2013-05-31; First posted 2013-06-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-12-15

CONDITIONS: Nicotine Dependence
Keywords: Smoking Cessation; fMRI; e-Cigarettes; Natural History
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ex-smokers: former smokers who have quit
- never smokers/vapers: never smoked/vaped nicotine
- non-treatment seeking smokers/vapers: smokers/vapers not interested in quitting nicotine
- Treatment seeking smokers/vapers: smokers/vapers interested in quitting nicotine

SUMMARY:
Background:

- Smoking is a difficult habit to quit, and some people find it more difficult to quit than others do. Nicotine is the substance in cigarettes that makes smoking so addictive. Nicotine changes some patterns of brain activity, and smokers have differences in brain activity when compared to non-smokers. Some genes make it more likely that a person will become addicted to smoking. Researchers want to study how nicotine interacts with genes and brain activity. This may help develop better treatments to help people quit smoking.

Objectives:

- To develop a test of nicotine dependence, using brain activity and genetic analysis, which may be useful in predicting success in smoking cessation and in the development of new smoking cessation treatment targets.

Eligibility:

* Main group: Current smokers between 18 and 55 years of age who are seeking treatment to quit.
* Comparison group: Current smokers between 18 and 55 years of age who are not seeking to quit.
* Comparison group: Healthy former smokers between 18 and 55 years of age.
* Comparison group: Healthy nonsmoking volunteers between 18 and 55 years of age.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be collected.
* The three comparison groups will have one magnetic resonance imaging (MRI) scan session. They will have tests of thinking, concentration, and memory both inside the scanner, and while sitting in front of a computer.
* Current smokers who are trying to quit must be willing to undergo a course of nicotine treatment that includes weekly counseling (for 12 weeks) and e-cigarettes. Participants will attempt smoking abstinence and will have a total of 6 MRI scanning sessions. They will do thinking, concentration, and memory tasks inside and outside of the scanner.
* For smokers, the first scanning session will take place before they attempt to quit. This will be a baseline scan. The second scanning session will take place 48 hours after having their last real cigarette. After this scan, they will use electronic cigarettes to help quit their habit.
* After using e-cigarettes for two weeks, smokers will have a third scan session.. They will then gradually taper their use of the electronic cigarettes over the course of three weeks, at which point they will be nicotine abstinent.
* After about 5 weeks of abstinence, they will have the fourth scan. The fifth scan will be approximately 6 months after start of the study, and the final scan will take place at about 1 year from the study start.
* Smokers will continue to receive support on quitting smoking until the study ends at about 1 year.

DETAILED DESCRIPTION:
Objective: To develop a neuroimaging/genetic/epigenetic biomarker of nicotine dependence severity that may be useful in predicting success in smoking cessation and in development of new smoking cessation treatment targets. Further, by evaluating those who vape nicotine, findings will determine whether biomarkers differ between those who smoke or vape, allowing for the development of cessation

strategies that relate to preferred nicotine delivery.

Study population: Four groups will be studied: target group of treatment seeking smokers/vapers; nontreatment seeking current smokers/vapers; never smokers/never vapers and former smokers. We estimate that we will need n=50/subgroup completers to have sufficient power to develop the brain/genetics biomarkers.

Design: This study consists of a 4 group between/within subject design. The experimental group will proceed in 4 phases: Baseline (scan 1), peak withdrawal (scan 2), stable on nicotine replacement (scan 3), and complete abstinence (scans 4-6). Counseling will start after the first scan session and will generally continue weekly until scan 4 (about 12 weeks). After scan 4, therapeutic support will be

provided at least monthly via phone until completion of the protocol. The non-treatment seeker comparison group will be scanned twice; at baseline (scan 1) and at peak withdrawal (scan 2). Each of the non-nicotine user comparison groups (non-nicotine users and Ex-smokers) will be scanned only at baseline (scan 1). Genetic and epigenetic markers will be obtained in all groups.

Outcome measures: Network and multivariate pattern analysis, behavior on a decision making task and task based and resting state blood oxygen level-dependent (BOLD) activation in neural circuits relevant to nicotine addiction during fMRI scanning. Secondary outcomes include BOLD response comparisons between nicotine replacement and typical nicotine use and genetic markers of nicotine addiction and relapse susceptibility.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants must:

1. Be between the ages of 18-60. Assessment tool(s): Edinburgh Handedness Inventory. Although left-handed individuals will not be excluded, we will track handedness. Justification: Some of the neural processes assessed in this protocol may be lateralized in the brain. In order to assess potential variance, participants handedness will be documented.
2. Be in good health. Justification: Many illnesses may alter fMRI signals as well as cognitive processes and neural functioning. Assessment tool(s): Participants will provide a brief health history during phone screening, and undergo a medical history and physical examination with a qualified IRP clinician.
3. Be free of active DSM-IV dependence, on alcohol or any drug except nicotine. Past active dependence is acceptable provided it is at least two years in the past. Those with past dependence on substances other than alcohol or marijuana may not have any current use (past 6 months) of the substance on which they were dependent. Individuals with past dependence on either alcohol or marijuana who report current use of the previously dependent substance may be included, provided they do not currently meet any criteria for dependence, with the exception of tolerance. MAI may exclude on a case-by-case basis for heavy alcohol or drug use not meeting dependence criteria but likely to interfere with data quality. Justification: Dependence on other substances (drugs or alcohol) may result in unique CNS deficits that could confound results and introduce excessive variance. Assessment tool(s): The SCID and/or the Mini International Neuropsychiatric Interview (M.I.N.I) and clinical substance abuse/dependence assessment. While recreational/intermittent use of alcohol and/or marijuana will be tolerated in all participant groups, individuals will be excluded if they meet current or recent (within 2 years) DSM-IV diagnostic criteria for dependence on any substances. A positive drug test for marijuana will not be exclusionary as long as participants have not used in the 24hrs preceding the imaging visits. In the event of a positive drug test for marijuana, self-reports of current marijuana use will be used to differentiate intermittent/infrequent from chronic/frequent users.
4. Be able to abstain from alcohol 24hrs before each of the imaging sessions and able to abstain from caffeine 24hrs before each session. Justification: Alcohol and caffeine modulate neural functioning in a way that would complicate data interpretation. Assessment tool(s): Self-report and breathalyzer.
5. For the treatment and non-treatment seeking groups, must have a urine cotinine level corresponding to smoker/nicotine user status for the specific test being used (typically corresponding to a urine cotinine above about 200 ng/ml) and have been smoking or vaping consistently for at least the past year (excluding quit attempts). Based on the correlation between self-reported cpd/FTND and urine cotinine levels [85a, 85b], a single inclusion criterion will be easier to manage and provide adequate characterization of nicotine dependent participants. Urine cotinine level provides a biomarker that does not rely on self-report/memory. Quit attempts will be assessed via clinical interview and judgment. Justification: The present protocol is interested in neurobiological mechanisms that underlie nicotine dependence-induced plasticity and is thus contingent on the presence of nicotine dependence. Assessment tool(s): Self-report, commercial urine cotinine test corresponding to smoker/nicotine user status for the specific test being used, typically corresponding to a urine cotinine above about 200 ng/ml.
6. For the treatment and non-treatment seeking groups, must be willing to attempt an acute abstinence period lasting approximately 48 hours.
7. For the treatment seeking group, be actively seeking treatment for nicotine cessation and willing to engage in 12-weeks of treatment involving weekly counseling sessions, as well as follow-up imaging and behavioral assessments following treatment onset.
8. For the ex-smoker group, must have smoked approximately 8 or more cigarettes per day for at least 1 year, and have remained abstinent continuously for at least the last 12 months. Justification: While serum cotinine level has been shown to be a more accurate measure of cigarette smoking than CPD [85c], it is impossible in the current design to collect retroactive serum cotinine levels from exsmokers. Instead, CPD must be equated with the urine cotinine levels of current treatment and nontreatment seeking groups. The low-end cotinine level for the inclusion of smokers/vapers in this protocol is about 200 ng/mL. In adult smokers, a nicotine intake of approximately 1 mg can be estimated from a blood cotinine level of 12.5 ng/mL) [85d]. Thus, to have achieved a blood cotinine level of 200ng/mL, ex-smokers would have to self-report consumption of 16 mg of nicotine per day which equates to approximately 8 CPD (0.36-2.62 mg nicotine yield per cigarette [85e]. Given these calculations, the inclusion criterion for the ex-smoker group has been lowered to 8 CPD. Assessment tool(s): Self-report, commercial urine cotinine test corresponding to non-smoker status for the specific test being used, typically corresponding to a urine cotinine under about 20 ng/ml, CO < 6.
9. For the non-smoking/vaping control group, less than 20 times of lifetime use of nicotine containing products and vaping of non-nicotine containing products, none in past year and no history of daily nicotine use. Justification: Minimal nicotine exposure in the control group is required to assess differences between controls and the nicotine groups. Assessment tool(s): Self-report, commercial urine cotinine test corresponding to non-smoker status for the specific test being used, typically corresponding to a urine cotinine under about 20 ng/ml, CO < 6.

EXCLUSION CRITERIA:

3.3 Exclusion criteria:

Participants will be excluded if they:

1. are not suitable to undergo an fMRI experiment due to certain implanted devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology, or claustrophobia. Justification: MR scanning is one of the primary measurement tools used in the protocol. Assessment tool(s): Prospective participants will fill out an MRI screening questionnaire and undergo an interview with an MR technologist. Questions concerning suitability for scanning will be referred to the MR Medical Safety Officer. Prospective participants will be questioned about symptoms of claustrophobia and placed in the mock scanner during their first visit to assess for possible difficulty tolerating the confinement of the scanner and for ability to fit into the scanner.
2. have coagulopathies, history of, current superficial, or deep vein thrombosis, musculoskeletal

   abnormalities restricting an individual s ability to lie flat for extended periods of time. Justification: MR scanning sessions require participants to lie flat on their backs and remain perfectly still for approximately two hours. Therefore, conditions that would make that difficult (e.g. chronic back pain, significant scoliosis) or dangerous (e.g. familial hypercoagulability syndrome, history of thrombosis) will be exclusionary. Assessment tool(s): History and physical examination by a qualified IRP clinician, supplemented with a trial of lying in the mock scanner to assess comfort issues.
3. have HIV or Syphilis. Justification: HIV and Syphilis both can have central nervous system (CNS) sequelae, thus introducing unnecessary variability into the data. Assessment tool(s): Oral HIV blood test if oral test is + and STS+ without adequate prior treatment
4. regularly use any prescription (e.g., benzodiazepines, antipsychotics, anticonvulsants, barbiturates), over-the-counter (e.g., cold medicine) or herbal medication (e.g., Kava, Gingko biloba, St. John s wort) that may alter CNS function, cardiovascular function, or neuronal-vascular coupling. Antidepressant use will be allowed if an individual is on a stable dose of an SSRI or SNRI for ~6 weeks. As needed, benzodiazepine use is also allowed, but the individual must test negative for benzodiazepines on the drug screen. Justification: The use of some medications may alter the fMRI signal and/or neural functions of interest in the current study. Consistent antidepressant use or infrequent use of benzodiazepines is unlikely to drive study-related changes in brain function. Allowing such medication use will also make it possible to study nicotine dependent individuals who continue to smoke despite receiving treatment for a mood disorder. Assessment tool(s): History and comprehensive urine drug screening to detect antidepressants, benzodiazepines, antipsychotics, anticonvulsants, and barbiturates.
5. have any current neurological illnesses including, but not limited to, seizure disorders, frequent migraines or on prophylaxis, multiple sclerosis, movement disorders, history of significant head trauma, or CNS tumor. Justification: Neurological diseases alter CNS function and, possibly, the neuronalvascular coupling that forms the basis of the fMRI signal. Assessment tool(s): History and physical examination by a qualified IRP clinician, urine drug screening for anticonvulsants not disclosed by history. History of head trauma with loss of consciousness of more than 30 minutes or with postconcussive sequelae lasting more than two days, regardless of loss of consciousness, will be exclusionary. The MAI who will also retain discretion to exclude based on a history of neurological illness that may compromise data integrity.
6. Have current major psychiatric disorders to include, but not limited to psychotic disorders, or substance-induced psychiatric disorders, or risk of suicide or currently on antipsychotic medication treatment. Individuals with current major depressive disorder (MDD) and related anxiety will be allowed if currently stable, as assessed by the MAI. The MAI will reserve the right to exclude on the basis of psychiatric history not explicitly described in this criterion. Justification: Psychiatric disorders involve the central neural system (CNS) and, therefore, can be expected to alter the fMRI measures being used in this study. However, mood disorders such as MDD are highly comorbid with nicotine dependence. Including this population will generate results that are more representative of nicotine dependent individuals. Assessment tool(s): Computerized SCID or M.I.N.I., Beck Depression Inventory, Beck Anxiety Inventory, Adult ADHD Self-Report Scales and clinical interview confirmation by clinician.
7. Are cognitively impaired or learning disabled. Justification: Cognitive impairment and learning disabilities may be associated with altered brain functioning in regions recruited during laboratory task performance. Cognitive impairment may affect one s ability to give informed consent. Assessment tool(s): History examination and validated IQ test, such as the Wechsler Abbreviated Scale of Intelligence (WASI) or Shipley-2. IQ estimate must be 80 or over.
8. have significant cardiovascular, cerebrovascular, or respiratory conditions. Justification: Such conditions may alter blood flow, the fMRI signal and other autonomic signals, and increase risks associated with nicotine patch and/or e-cigarette use. Assessment tool(s): History and physical exam, including 12-lead EKG.
9. have any other major medical condition that in the view of the investigators would compromise the safety of an individual during participation. Justification: Many illnesses not explicitly covered here may increase risk or alter important outcome measures. Assessment tool(s): History and physical examination by a qualified IRP clinician and CBC, urinalysis, NIDA chemistry panel (liver function tests, electrolytes, kidney function). The following lab values will result in exclusion from the study:

   i. Hemoglobin < 10 g/dl

   ii. White Blood Cell Count < 2400/ l

   iii. Liver Function Tests > 3X normal

   iv. Serum glucose > 200 mg/dl

   v. Urine protein > 2+

   vi. Serum creatinine > 2 mg/dl

   vii. Estimated creatinine clearance <60ml/min

   The MAI will retain discretion to exclude based on less extreme lab results. After the screening process has been completed, the MAI will take into account all data collected in order to decide if there is an existing medical illness that would compromise participation in this research.
10. are pregnant, planning to become pregnant, or breastfeeding. Females are instructed in the consent to use effective forms of birth control during the study period. Justification: study procedures and drugs used in the current protocol may complicate pregnancy or be transferred to nursing children. Assessment tool(s): Urine and/or serum pregnancy tests, and clinical interview. Urine pregnancy tests will also be conducted at the beginning of each imaging visit.
11. Are non-English speaking. Justification: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify, given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing MRI procedures. The inability to effectively communicate MRI safety procedures in a language other than English could compromise the safety of non-English speaking participants. Assessment tool(s): self-report....

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: No preferences in participant recruitment will be made on the bases of gender, race, or ethnic background. Efforts will be made to avoid participant distribution bias such that if skewing is noted, subjects in the over-represented group may temporarily be excluded from the study until additional participates from under-represented groups can be established. Efforts will be made to include minorities in proportion to their presence in the local population. The major metropolitan Baltimore area (Baltimore City, Baltimore County, Anne Arundel County, Howard County) consists of 64% White, 32% Black or African American, 3% Asian, 0.3% American Indian and Alaska Native, 0.04% Native Hawaiian and Other Pacific Islander and 0.8% some other race (http://www.census.gov/ ). Of this population (any race), 2% are Hispanic or Latino.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2013-11-06 (Actual); Primary Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Change in BOLD signal and functional connectivity related to task parameters, between drug conditions (i.e. on and off nicotine) and between groups | each scan visit
  1) Change in BOLD signal and functional connectivity related to task parameters, between drug conditions (i.e. on and off nicotine) and between groups: will provide important insight into the neurobiological mechanisms underlying acute and chronic nicotine withdrawal, in particular those related to anhedonia, negative affect, cognitive control and impulsive decision making.
Genetic and epigenetic data | each scan visit
  2) Genetic and epigenetic data. These data will be included into the network and pattern classification models discussed above as features in the classifier. They will also be used as regressors, covariates or dichotomous variable in the above BOLD task analysis.
Resting state MRI at follow-up | each scan visit
  3) Resting state MRI at follow-up. Resting state MRI will be assessed between- and within- groups as a function of relapse status and time since last treatment visit at each of the follow-up time-points (4 weeks, 3, 6 and 12 months). These data will be entered into the network and pattern classification models discussed above. This will allow us to address the following questions:i. What characteristics of rsFC are associated with treatment success (vs. failure)? ii. Are there characteristics of rsFC that vary as a function of time post-treatment in successfully abstinent individuals?
Behavioral performance on each task | each scan visit
  4) Behavioral performance on each of the tasks assessing working memory, attention, processing speed, inhibitory control processes, cognitive control, reward responsiveness, amygdala, striatal, and impulsive decision making (e.g., reaction time, error rate, hit rate, reward bias): will provide task-related parameters necessary for analysis of BOLD and resting state data. Performance data will function as a secondary outcome by providing behavioral validation of acute and chronic nicotine withdrawal effects.
Self-reported craving, withdrawal symptoms & mood/affect | each scan visit
  5) Self-reported craving, withdrawal symptoms and mood/affect: will be employed as regressors in the analysis of task and resting BOLD data. They will also provide the primary means of validating the acute nicotine withdrawal manipulation.
Smoking status at 4wks, 3, 6 and 12 months. | each scan visit
  6) Smoking status at 4 weeks, 3, 6 and 12 months: Smoking status (relapse vs. abstinent) at each of the follow-up time points will be based on 7-day point prevalence defined as no smoking (not even a puff) or use of any tobacco products for the past 7 days. This is a standard method of assessing abstinence and dichotomizing relapse status at follow-up. Whenever abstinence at follow-up is assessed in-person, self-reported abstinence will be corroborated with breath COand urine cotinine levels.

SECONDARY OUTCOMES:
2) Structural MRI and DTI data | each visit
  2) Structural MRI and DTI data
1) Ratings and scores on self-report characterization measures | each visit
  1) Ratings and scores on self report characterization measures

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Janes, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share IPD for this protocol; however, plans have not yet been finalized. We have not yet finalized decisions on types of supporting information that will be shared, IPD Sharing Time Frame, or IPD Sharing Access Criteria. Data will be stripped of identifiers prior to release for sharing. De-identified data may be shared with properly administered databases and/or with collaborators with whom proper data sharing agreements are in place (we will set-up proper data sharing agreements once a plan is determined).